CLINICAL TRIAL: NCT03064334
Title: Patients' Views on Outcomes Following Total Knee Arthroplasty: a Focus-group Study
Status: Completed | Type: Observational
Sponsor: University of Salford (Other)
Collaborators: Stockport NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Bodor Bin sheeha, PhD student, University of Salford
Other Study IDs: qualitative
Record Dates: First submitted 2017-02-15; First posted 2017-02-27 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one medium of focus groups: The present study aims to understand patient experiences and outcomes post- Total Knee Arthroplasty(TKA). Therefore, a qualitative approach will be most appropriate to facilitate the collection of in-depth experiences and perceptions of patients post-TKA.
  The medium of focus groups (with 8-10 patients) is preferred to allow a group of patients to share their perceptions and experiences post-surgery, with sufficient quantity and diversity of views while balancing the facilitator's ability to manage all patients' participation for 90-120 minutes (Bloor, 2006).
  Interventions: Procedure: Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — surgical knee joints Arthroplasty
  Other Names: Total Knee Replacement surgery

SUMMARY:
In order to assess patients' concerns and other quality of life aspects, post-total knee arthroplasty (TKA) requires further assessment tools, more than controlled experiments testing defined isolated variables. Qualitative research offers useful methods to explicate the complexity and deeper meaning of patient experiences and outcomes post-TKA. Qualitative methods facilitate the collection of in-depth experiences and perceptions from individuals about a specific phenomenon which, in this case, is outcomes post-TKA. Specifically, a phenomenological approach allows for the collection of diverse and unique patient experiences and outcomes post-TKA .

The focus of this project is using focus groups to explore poorly understood areas, such as outcomes and experiences post-TKA, in order to generate useful findings and hypotheses.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a major cause of disability around the world; it is the most common chronic condition in primary care in the UK. By 2030 it is predicted to be the greatest cause of disability in the general population . An effective end-stage treatment for knee OA is knee-replacement surgery, which was first done in the 1970s and 1980s.

In England and Wales, the number of knee-replacement procedures recorded by the National Joint Registry in 2013 was 91,703, which represents an increase of 0.9 % over 2012. The data analysis by the National Joint Registry and the Office of National Statistics suggests that, by 2030, primary Total Knee Arthroplasty (TKA) will increase by 117% from the 2012 level. Subsequently, TKA revision surgeries are expected to increase incrementally by 332%. There is a similar estimation of demand for revision TKA surgeries in the United States; by 2030, they are expected to rise by 601% from the 2005 level. The United States estimation of primary TKA is for growth of 673% from the 2005 level, which is similar to England and Wales's upper-limit projections .

Post-TKA, 75-85% of patients report satisfaction with surgery outcomes, while the remaining 15-25% are dissatisfied .Total knee arthroplasty's success has traditionally been evaluated from the surgeon's perspective, e.g. the presence of surgical complications or implant survival. This is gradually changing to involve the patient in measuring health outcomes and decision-making processes. Patient-reported outcome measures (PROMs) have evolved to explore patient perspectives by monitoring the quality of care in health organizations and conducting clinical trial outcomes.

More than half of patients' early concerns post-total knee arthroplasty (TKA) are not considered in commonly used patient-reported outcome measures . This may support current medical outcomes evaluation post-TKA having implications that differ from the patient perspective. This may be explained by the dissatisfaction of some patients post-TKA. So, being more sensitive to patient experience assessment methods is required, rather than profession-driven tools.

Patients' experiences and their perceptions of current outcome measurements post-TKA are poorly understood. In order to explore this area qualitative methods are appropriate, as they facilitate the collection of in-depth experiences and perceptions of individuals about a specific phenomenon which, in this case, is outcomes post TKA. Specifically, a phenomenological approach allows for the collection of diverse and unique patient experiences and outcomes post-TKA.

A focus group is useful for exploring poorly understood areas, such as outcomes and experiences post-TKA, in order to generate possible findings or hypotheses. It has advantages over one-to-one interviews as the interaction among group members provides an extra dimension to gather data and a wider degree of spontaneity in the patient views expressed, in contrast to one-to-one interviews where the interaction is limited to that between patients and researcher and depends on patient responses. Interaction in a group setting allows patients to refine their views in light of others' views and facilitates further spontaneous expression. Support for the feelings of other group members with similar experiences encourages less verbal individuals to contribute more than in one-to-one interviews.

Only three previous studies have used focus-group methods to explore patient experiences post-TKA. Studies by Westby et al. (2010) and Van Egmond et al. (2015) combined the results of patient experiences post-total knee arthroplasty and post-total hip arthroplasty, which does not support accuracy as those patient groups encounter different problems. The third study, by Zacharia et al. (2016), assessed outcomes at least three years post-TKA in a limited age range of 60-65 years for manual labourers of low and medium socioeconomic status. An appropriate well-structured methodology is required to explore patient experiences and outcomes post-TKA, with clear sampling and population criteria to facilitate the possible correlation of findings.

To the best of our knowledge, no study has explored patient experiences and outcomes post-TKA using focus-group discussions one year after surgery to explore whether there are factors that might help us to understand why some patient medical outcome measurements were good but they were not satisfied, or vice versa. Exploration of potential barriers to functional recovery may support future modifications that might improve outcomes post-TKA.

Project objectives

* To gain an in-depth understanding of experiences and perceptions of patients about outcomes post-TKA and to explore whether there are factors that might help us understand why some patients' medical outcome measurements were good but they were not satisfied, or vice versa.
* To gain insights into potential barriers to good functional recovery.
* To identify what modifications can be made to improve future outcomes post-TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone primary unilateral total knee arthroplasty within the last year.
* Maximum post-operative achievement is between one and two years.
* Patients can read and understand English, non-English speaking patients will be excluded from the study to avoid any language barrier.
* Purposive sampling will be used to recruit the most relevant patients to answer the research questions such as;
* mixed genders to explore gender-experience differences.
* mixed work and retired to explore return to work barriers
* patients with family support and patients living alone to explore the value of family support or home-care services
* mixed educational levels to explore educational background effects.

So there will be no age, gender, social, work status or educational level limitations (Schwandt, 2001)

Exclusion Criteria:

There are possible complications or they present with other pathological conditions that might change recovery progression, they will be excluded to minimize confounding factors and their effects on patients' experiences and outcomes, such as:

* They have undergone bilateral knee arthroplasty, unilateral knee revision surgery, post-traumatic or unicompartmental knee replacement.
* They cannot read and understand English.
* Their function is limited due to musculoskeletal involvements other than unilateral knee osteoarthritis.
* They have been diagnosed with uncontrolled diabetes mellitus or blood pressure.
* Post-TKR they are in pathological groups, such as having neurological disorders (stroke, Parkinson's disease etc.), haemophilia or psychological pathologies.
* They are morbidly obese and have a body mass index (BMI) greater than 40.
* They have advanced osteoporosis or some other unstable chronic disease.
* They have been diagnosed with peripheral vascular disease or an uncontrolled cardiac disease.
* They present with major postoperative complications, such as infection, fracture, acute myocardial infarction, stroke, pulmonary embolism or deep-vein thrombosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participants will be recruited at Stepping Hill Hospital. Sample criteria require will be clarified for all three orthopaedic surgeons at the hospital. Any patients attending for a one-year follow-up visit who are willing to participate in a focus-group study will be included in a research-patients list. A participant information sheet and an informed consent form will be sent via Royal Mail or email to each participant four weeks before the study to allow participants to consider their involvement in the study and have the time to decide whether or not to contribute. They will be able to change their minds on the day should they wish to do so.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Medium focus groups discussion to explore the patients experiance and functional recovery post -TKA. | 60 -70 minute of total 120 minute of focus group discussion.
  Qualitative methods in term of medium focus groups discussion will be used to explore the patients perceptions and experiences post-surgery. The focus groups will be facilitated by a focus-group expert and the researcher using open-ended questions in order to prompt free discussion to explore their experience and barrier post-TKA. All topics and questions covered will be suitable to discuss in a semi-public setting. All discussions will be recorded using electronic methods, in addition to field notes taken by both facilitator and researcher.
  Discussion guide: How was experience of Total Knee Arthroplasty (TKA), Functional improvements after TKA, What modifications have been made to compensate for that, What are the barrier, In the course of routine activities did the patients need help, Did the patients need family support, Were patients able return to work after TKA, (if not, why? what are the barriers

SECONDARY OUTCOMES:
Medium focus groups discussion to explore the quality of health service provide post -TKA | 40 -50 minute of total 120 minute of focus group discussion.
  The secondary outcome from the focus group discussion will Evaluate the health service quality using the following questions; How did the patients feel about the surgery now? Did patients satisfy all their expectations, Did they receive sufficient information and explanation about surgery and expectations in advance from the health team, Was that sufficient for what they needed to know before surgery, Do patient think that has affected their satisfaction after surgery, Have they received physiotherapy post-surgery. For how long How many sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Richard Professor Jones, Study Director — Director of the Salford University Gait Laboratory
Locations (1):
- Stockport NHS Foundation Trust, Stockport, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attride-Stirling, J. (2001). Thematic networks: an analytic tool for qualitative research. Qualitative Research, 1(3), 385-405. doi:10.1177/146879410100100307
- [Background] Beaton DE, Clark JP. Qualitative research: a review of methods with use of examples from the total knee replacement literature. J Bone Joint Surg Am. 2009 May;91 Suppl 3:107-12. doi: 10.2106/JBJS.H.01631. PMID 19411508
- [Background] Bloor, M., and Wood, F. (2006). Keywords in Qualitative Methods. A Vocabulary of Research Methods. London: SAGE Publications Ltd.
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Hossain FS, Konan S, Patel S, Rodriguez-Merchan EC, Haddad FS. The assessment of outcome after total knee arthroplasty: are we there yet? Bone Joint J. 2015 Jan;97-B(1):3-9. doi: 10.1302/0301-620X.97B1.34434. PMID 25568406
- [Background] Jagger, C., Matthews, R., Spiers, N., Brayne, C., Comas - Herrera, A., Robinson, T., . . . Croft, P. (2006). Compression or expansion of disability?: forecasting future disability levels under changing patterns of diseases: King's Fund.
- [Background] Kitzinger J. Qualitative research. Introducing focus groups. BMJ. 1995 Jul 29;311(7000):299-302. doi: 10.1136/bmj.311.7000.299. PMID 7633241
- [Background] Klit J, Jacobsen S, Rosenlund S, Sonne-Holm S, Troelsen A. Total knee arthroplasty in younger patients evaluated by alternative outcome measures. J Arthroplasty. 2014 May;29(5):912-7. doi: 10.1016/j.arth.2013.09.035. Epub 2013 Oct 1. PMID 24269097
- [Background] Lehoux P, Poland B, Daudelin G. Focus group research and "the patient's view". Soc Sci Med. 2006 Oct;63(8):2091-104. doi: 10.1016/j.socscimed.2006.05.016. Epub 2006 Jun 23. PMID 16797811
- [Background] Ong BN, Richardson JC. The contribution of qualitative approaches to musculoskeletal research. Rheumatology (Oxford). 2006 Apr;45(4):369-70. doi: 10.1093/rheumatology/kel022. Epub 2006 Jan 25. No abstract available. PMID 16436487
- [Background] Palomba, C. A., & Banta, T. W. (1999). Assessment essentials : planning, implementing, and improving assessment in higher education. San Francisco: Jossey-Bass Publishers.
- [Background] Patel A, Pavlou G, Mujica-Mota RE, Toms AD. The epidemiology of revision total knee and hip arthroplasty in England and Wales: a comparative analysis with projections for the United States. A study using the National Joint Registry dataset. Bone Joint J. 2015 Aug;97-B(8):1076-81. doi: 10.1302/0301-620X.97B8.35170. PMID 26224824
- [Background] Rastogi R, Davis AM, Chesworth BM. A cross-sectional look at patient concerns in the first six weeks following primary total knee arthroplasty. Health Qual Life Outcomes. 2007 Aug 1;5:48. doi: 10.1186/1477-7525-5-48. PMID 17678532
- [Background] Sandelowski M. Sample size in qualitative research. Res Nurs Health. 1995 Apr;18(2):179-83. doi: 10.1002/nur.4770180211. PMID 7899572
- [Background] Schwandt, T. (2001). Dictionary of Qualitative Inquiry: Thousand Oaks Ca: Sage.
- [Background] Sim, J., & Snell, J. (1996). Focus groups in physiotherapy evaluation and research. Physiotherapy, 82(3), 189-198.
- [Background] van Egmond JC, Verburg H, Vehmeijer SB, Mathijssen NM. Early follow-up after primary total knee and total hip arthroplasty with rapid recovery : Focus groups. Acta Orthop Belg. 2015 Sep;81(3):447-53. PMID 26435240
- [Background] Westby MD, Backman CL. Patient and health professional views on rehabilitation practices and outcomes following total hip and knee arthroplasty for osteoarthritis:a focus group study. BMC Health Serv Res. 2010 May 11;10:119. doi: 10.1186/1472-6963-10-119. PMID 20459834
- [Background] Williams DP, Blakey CM, Hadfield SG, Murray DW, Price AJ, Field RE. Long-term trends in the Oxford knee score following total knee replacement. Bone Joint J. 2013 Jan;95-B(1):45-51. doi: 10.1302/0301-620X.95B1.28573. PMID 23307672
- [Background] Zacharia B, Paul M, Thanveeruddin Sherule M. Patient-based outcome analysis is important to determine the success of total knee arthroplasty: result of a focus group discussion. Med Devices (Auckl). 2016 May 23;9:125-30. doi: 10.2147/MDER.S97094. eCollection 2016. PMID 27284268